CLINICAL TRIAL: NCT00030121
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Evaluation of the Safety and Efficacy of Carperitide Infusion in Patients With ARDS
Brief Title: Carperitide in Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suntory Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPI-001
Record Dates: First submitted 2002-01-31; First posted 2002-02-01 (Estimated); Last update posted 2008-02-20 (Estimated); Status verified 2008-02

CONDITIONS: Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress; Acute Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

INTERVENTIONS:
Drug: recombinant human atrial natriuretic polypeptide

SUMMARY:
The purpose of this study is to determine whether Carperitide is safe and effective in the management of Acute Respiratory Distress Syndrome (ARDS).

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS is a severe form of acute lung injury. ARDS is characterized by an increase in pulmonary vascular permeability resulting from a non-cardiogenic cause, leading to an increased vascular water volume, pulmonary inflammation, and severe hypoxemia. Conventional therapy for ARDS is primarily respiratory management by mechanical ventilation using positive end-expiratory pressure (PEEP). Mechanical ventilation is the major management concern in patients with ARDS, due to its higher risk of infections and morbidity. Treatment with Carperitide may reduce time on the ventilator by reducing pulmonary edema and by improving gas exchange. The results of Carperitide studies in animals and humans support the idea that the hormone will be effective in managing the acute pulmonary complications and hypoxemia seen in ARDS.

ELIGIBILITY:
Inclusion:

In order to participate in the study, patients must:

* be 18 years or older
* have an acceptable PF ratio
* have adequate fluid volume
* be intubated less than 7 days

Exclusion:

In order to participate in the study, patients must not meet any of the following criteria:

* be moribund
* be immunocompromised
* have pneumonia (caused by Pneumocystis carinii)
* have recieved another investigational drug or device within the last 30 days
* have a Do not Resuscitate order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12